CLINICAL TRIAL: NCT05229289
Title: Efficacy and Safety of Fecal Microbiota Transplant for Secondary Prophylaxis of Hepatic Encephalopathy: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Fecal Microbiota Transplant for Secondary Prophylaxis of Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS- Cirrhosis-40
Record Dates: First submitted 2021-12-24; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-12

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT along with SMT (Experimental): FMT + Standard medical therapy (SMT):
  Lactulose (Titrated to 2-3 soft bowel movements per day) Oral LOLA can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Oral BCAAs can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Diet Daily energy intakes of 35-40 kcal/kg ideal body weight Daily protein intake 1.2-1.5 g/kg/day Small meals or liquid nutritional supplements evenly distributed throughout the day Oral BCAA supplementation in patient's intolerant of dietary protein (to allow recommended nitrogen intake to be achieved and maintained)
  Interventions: Other: Standard Medical Treatment; Other: Fecal Microbiota Transplant
- Standard Medical Treatment (Active Comparator): Standard medical therapy (SMT):
  Lactulose (Titrated to 2-3 soft bowel movements per day) Oral LOLA can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Oral BCAAs can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Diet Daily energy intakes of 35-40 kcal/kg ideal body weight Daily protein intake 1.2-1.5 g/kg/day Small meals or liquid nutritional supplements evenly distributed throughout the day Oral BCAA supplementation in patient's intolerant of dietary protein (to allow recommended nitrogen intake to be achieved and maintained)
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Other: Standard Medical Treatment — Standard medical therapy (SMT):
  Lactulose (Titrated to 2-3 soft bowel movements per day) Oral LOLA can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Oral BCAAs can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Diet Daily energy intakes of 35-40 kcal/kg ideal body weight Daily protein intake 1.2-1.5 g/kg/day Small meals or liquid nutritional supplements evenly distributed throughout the day Oral BCAA supplementation in patient's intolerant of dietary protein (to allow recommended nitrogen intake to be achieved and maintained)
Other: Fecal Microbiota Transplant — Fecal Microbiota Transplant
  Arms: FMT along with SMT

SUMMARY:
Despite standard of care, the recurrence of hepatic encephalopathy remains the primary cause for readmissions in individuals with cirrhosis. Patients with cirrhosis have disturbed gut microbiota, which is exacerbated by repeated antibiotic usage. FMT is a promising therapy to restore a healthy microbiota. FMT causes change in composition of gut microbiota which will lead to increase in commensal bacterial diversity which will increase colonization resistance to pathogenic bacteria and thereby decrease the bacterial overgrowth. Healthy bacteria also increase the SCFA production in colon with is and nutrient for endothelial cells and thereby protect the endothelial integrity and decreases bacterial translocation and endotoxemia. Current standard of care mainly focuses on the treatment of precipitating factors of the HE. The goal of our open-label, randomised clinical trial is to evaluate the safety, efficacy of addition of FMT to SOC in preventing subsequent episodes of hepatic encephalopathy.

DETAILED DESCRIPTION:
Hypothesis Engraftment of healthy donor microbiota in cirrhotic patients with hepatic encephalopathy curtails dysbiosis which subsequently prevent further episodes of hepatic encephalopathy and thereby increasing the transplant free survival

AIM:-To study efficacy and safety of fecal microbiota transplantation in preventing recurrence of hepatic encephalopathy in patients with cirrhosis who have recovered from first episode of hepatic encephalopathy

Methodology Study population: All cirrhotic patients between 18 years to 70 years, who have recovered within 7 days from hepatic encephalopathy after hospitalization.

Study design: A Randomized Controlled Trial Study period: December 2021- December 2022 Sample size: 66 (44:22 cases in each group) Randomization: The randomization will be done in 2:1 ratio by block randomization method with block size of 6. The allocation concealment will be done by using SNOSE method.

There are no Indian studies (RCT) available for suggesting role of FMT in hepatic encephalopathy.

In the RCT by BAJAJ ET AL. HEPATOLOGY, December 2017, the incidence of HE in standard group was 60% (6/10) and 0%(0/10) in experimental group.

But this was and underpowered study and possibility of type 2 error is there. Assuming that there is 5% risk of development of HE in Experimental group (FMT with SMT) and 60% in SMT group with alpha 5%, power 90% with 2:1 allocation and considering 10% drop out rate, investigator decided to enroll 66 patients, 44 patients in experiential group and 22 patients in standard group

Intervention: This RCT will be conducted at ILBS New Delhi All cirrhotic patients between 18 years to 70 years, who have recently recovered from hepatic encephalopathy will be randomized into two groups.

Both groups will be given standard medical therapy,

Standard medical therapy (SMT):

Lactulose (Titrated to 2-3 soft bowel movements per day) Oral LOLA can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Oral BCAAs can be used as an alternative or additional agent to treat patients non-responsive to conventional therapy Diet Daily energy intakes of 35-40 kcal/kg ideal body weight Daily protein intake 1.2-1.5 g/kg/day Small meals or liquid nutritional supplements evenly distributed throughout the day Oral BCAA supplementation in patient's intolerant of dietary protein (to allow recommended nitrogen intake to be achieved and maintained) Group 1 will receive standard medical therapy only Group 2 will be given FMT along with SMT Healthy donor will be screen as per ILBS FMT proforma

Stool collection:

Donors will be supplied clean, sealable containers for collection and transport of stool. Containers will be labelled with the name, UHID and date/time of stool collection.

Collected stool will be immediately transferred to the laboratory facility for processing and used within 6 hours collection Stool sample from Healthy donor will be processed

Patient preparation:

Patients will have completed at least 3-day antibiotic course in hospital No antibiotics will be given 12 hours before administration of FMT however he will he/she will continue on SMT for HE (precipitating event, lactulose and rifaximin) No antibiotic or will be given for at least a day after instillation of FMT For administration of FMT, Endoscopy or fluoroscopy guided NJ tube will be placed Testing for Small intestinal bacterial overgrowth (SIBO) using breath test will be performed in a small set of patients (~30% of study population i.e 20 patients) Methods of FMT infusion. Three doses (30ml one dose) of FMT will be given via jejunal port of NJ/NG tube

The following data will be recorded for each patient:

Day 0: CBC, LFT, KFT, Ammonia, MELD, CTP, Sr Bile acid, Stool Microbiome and bile acid profile, IL-6 Cognitive Assessment: Overt HE - WHC, Covert HE- PHES and CFF At discharge: CBC, LFT, KFT, Ammonia, MELD, CTP, Sr Bile acid, Stool Microbiome and bile acid profile, IL-6, Cognitive Assessment: Over-WHC, Covert- PHES and CFF, Marker of neuroinflammation (IL-1β, OX-42)[Biobank], Urinary metabolomics {hippurate, formate, and reduced phenylacetylglutamine (PAG)}[Biobank] At 1 month: CBC, LFT, KFT, Ammonia, MELD, CTP, Sr Bile acid, Stool Microbiome and bile acid profile, IL-6, Cognitive Assessment: Over-WHC, Covert- PHES and CFF, Marker of neuroinflammation (IL-1β, OX-42)[Biobank], Urinary metabolomics {hippurate, formate, and reduced phenylacetylglutamine (PAG)}[Biobank] At 3 month: CBC, LFT, KFT, Ammonia, MELD, CTP, Sr Bile acid, Stool Microbiome and bile acid profile, IL-6, Cognitive Assessment: Over-WHC, Covert- PHES and CFF, Marker of neuroinflammation (IL-1β, OX-42)[Biobank], Urinary metabolomics {hippurate, formate, and reduced phenylacetylglutamine (PAG)}[Biobank] At 6 month: CBC, LFT, KFT, Ammonia, MELD, CTP, Sr Bile acid, Stool Microbiome and bile acid profile, IL-6, Cognitive Assessment: Over-WHC, Covert- PHES and CFF, Marker of neuroinflammation (IL-1β, OX-42)[Biobank], Urinary metabolomics {hippurate, formate, and reduced phenylacetylglutamine (PAG)}[Biobank] During follow up If any patient develops an episode of hepatic encephalopathy, he will be treated with standard medical therapy and after stabilization patient will be started on oral rifaximin 550 mg per day, and patient will be followed up till 6 months from day of FMT

Monitoring and assessment: All the parameters of the objective and also noted any adverse effects.

Adverse effects: Nausea, Vomiting, Fever with chills, dyspnea Stopping rule: If patient decided to withdraw from study Ethical issues in the study and plans to address these issues. None

ELIGIBILITY:
Inclusion Criteria:

- All cirrhotic patients between 18 years to 70 years, who have recovered within 7 days from hepatic encephalopathy after hospitalization

Exclusion Criteria:

1. Patient having hepatic encephalopathy after obvious precipitants (eg. diuretics, dehydration)
2. Patients on immunosuppressive medications
3. Active Infection (documented blood culture positive, Imaging diagnosis or SIRS>=1)
4. AKI (Defined as per KIDGO guidelines)
5. GI Bleed (In past 14 days)
6. Hepatocellular carcinoma
7. Patient with portosystemic shunt with size >10mm
8. Patients with previous TIPS or shunt surgery
9. Patients with significant comorbid illness such as heart, respiratory, or renal failure
10. Any neurologic diseases such as Alzheimer's disease, Parkinson's disease
11. Non hepatic metabolic encephalopathies
12. Not willing for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing an episode of hepatic encephalopathy within 6 months | 6 months

SECONDARY OUTCOMES:
Proportion of patients developing adverse event related to FMT within 6 months | 6 months
Number of Participants with Transplant free survival at day 28 | Day 28
Number of Participants with Transplant free survival at day 90 | Day 90
Number of Participants with Transplant free survival at day 180 | Day 180
Change in Ammonia level at day baseline, 28 days | 28 days
Change in Psychometric test/CFF pre and post FMT at day baseline, 28 days | 28 days
Change in Psychometric test/CFF pre and post FMT at day baseline,90 days | 90 days
Change in Ammonia level pre and post FMT at day baseline,90 days | 90 days
Change in Ammonia level pre and post FMT at day baseline, 180 days. | 180 days
Change in Psychometric test/CFF pre and post FMT at day baseline, 180 days. | 180 days
Change in inflammatory markers pre and post FMT at day baseline | 0 day
Change in inflammatory markers pre and post FMT at 28 days | 28 days
Change in inflammatory markers pre and post FMT at 90 days. | 90 days
Change in inflammatory markers pre and post FMT at 180 days. | 180 days
Change in urinary metabolomics pre and post FMT at baseline, 28 days | 28 days
Change in Stool microbiome and metabolomics pre and post FMT at baseline, 28 days | 28 days
Change in Stool microbiome and metabolomics pre and post FMT at baseline, 90 days | 90 days
Change in urinary metabolomics pre and post FMT at baseline, 90 days | 90 days
Change in urinary metabolomics pre and post FMT at baseline, 180 days | 180 days
Change in Stool microbiome and metabolomics pre and post FMT at baseline, 180 days | 180 days
Change in CTP score | 28 days
  Child-Turcotte-Pugh ranges from 5 to 15. 5 is good and 15 is worse.
Change in MELD score | 28 days
  Model for End Stage Liver Disease (MELD) score ranges from 6 to 40, 6 is good and 40 is worse.
Change in CTP score | 90 days
  Child-Turcotte-Pugh ranges from 5 to 15, 5 is good and 15 is worse
Change in MELD score | 90 days
  Model for End Stage Liver Disease (MELD) score ranges from 6 to 40, 6 is good and 40 is worse.
Change in CTP score | 180 days
  Child-Turcotte-Pugh ranges from 5 to 15, 5 is good and 15 is worse.
Change in MELD score | 180 days
  Model for End Stage Liver Disease (MELD) score ranges from 6 to 40, 6 is good and 40 is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No